CLINICAL TRIAL: NCT03349697
Title: Phyllantus Amarus for the Protection of Liver Health: A Randomized, Double Blind, Placebo Controlled Crossover Study
Brief Title: Phyllantus Amarus for the Protection of Liver Health
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biotropics Malaysia Berhad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BIOT1200
Record Dates: First submitted 2017-11-17; First posted 2017-11-21 (Actual); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Healthy
Keywords: Liver Health; Hangover; Herbal supplement; Liver function

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Product then Placebo (Experimental)
  Interventions: Dietary Supplement: Phyllantus amarus; Other: Placebo
- Placebo then Active Product (Experimental)
  Interventions: Dietary Supplement: Phyllantus amarus; Other: Placebo

INTERVENTIONS:
Dietary Supplement: Phyllantus amarus
Other: Placebo

SUMMARY:
This study is a randomized, double-blind, placebo controlled crossover study. The purpose of this study is to assess the ability of Phyllantus amarus to protect the liver against temporary stress including oxidative stress induced by alcohol consumption.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female 21-50 years of age, inclusive.
* Subject consumes at least 5 servings of alcohol per week on a regular basis.
* Minimum POMS score of 15.
* Access to a computer and internet
* Subject is willing to maintain his or her habitual food and beverage intake (other than substitution of study food for similar products) and physical activity patterns throughout the study period.
* Body mass index (BMI) between 20 and 30 kg/m2.
* Subject is willing and able to comply with the alcohol consumption requirements.
* Subjects willing to stay in the clinic for two overnight stays
* Judged by the Investigator to be in general good health on the basis of medical history.
* Subject understands the study procedures and signs forms providing informed consent to participate in the study and authorization for release of relevant protected health information to the study investigator.

Exclusion Criteria:

* Any Liver condition including Hepatitis, Fatty Liver, Liver Disease.
* Liver Function greater than three times the upper level limit of normal
* History or record of aggressive or violent behavior
* Any significant GI condition that would potentially interfere with the evaluation of the study product [e.g., Ulcerative Colitis or Crohn's Disease, inflammatory bowel disease, irritable bowel syndrome, Clinically significant Gastritis, history of upper GI bleed (bleeding ulcer), chronic constipation (defined as <3 bowel movements per week), history of frequent diarrhea, history of surgery for weight loss, gastroparesis, clinically important lactose intolerance].
* Clinically significant renal, hepatic, endocrine (including diabetes mellitus), cardiac, pulmonary, pancreatic, neurologic, or biliary disorder.
* Known allergy or sensitivity to any ingredients in the study products.
* Extreme dietary habits (e.g., vegan, Atkins Diet, etc.).
* Recent (within two weeks of visit 1, week -1) episode of acute gastrointestinal illness such as nausea, vomiting, or diarrhea.
* Uncontrolled hypertension (systolic blood pressure _160 mm Hg or diastolic blood pressure _100 mm Hg at visit 1, week -1).
* History or presence of cancer in the prior two years, except for non-melanoma skin cancer.
* Any major trauma or surgical event within three months of visit 1, week -1.
* Recent use of antibiotics (within 6 weeks).
* Females who are pregnant, lactating, planning to be pregnant during the study period.
* Recent history of (within 12 months) or strong potential for alcohol or substance abuse. Alcohol abuse will be defined as >14 drinks per week (1 drink =12 ounces beer, 5 ounces wine, or 1 ½ ounces distilled spirits).
* Participation in a clinical study with exposure to any non-registered drug product within 30 days prior.
* Individual has a condition the Investigator believes would interfere with his or her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results or put the person at undue risk
* Current active respiratory illness at the time of screening
* Any immune system disorders
* Subjects with a history of perforation of the stomach or intestines
* Subjects who have had gastric bypass surgery
* Untreated Hypothyroidism
* Subjects with active eating disorder including anorexia nervosa, bulimia, and/or obsessive compulsive eating disorders
* Spinal cord injuries

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2010-07-13 (Actual); Primary Completion 2010-10-16 (Actual); Study Completion 2010-10-16 (Actual)

PRIMARY OUTCOMES:
Compare the effect of Phyllantus versus placebo on HS CRP levels in blood | 26 days
Compare the effect of Phyllantus versus placebo on the inflammatory cytokines in blood | 26 days
Compare the effect of Phyllantus versus placebo on liver function levels in blood | 26 days
Compare the effect of Phyllantus versus placebo on glutatoine peroxidase (GSH-Px) in blood | 26 days

SECONDARY OUTCOMES:
Compare the effect of Phyllantus versus placebo on hangover severity score | 26 days
Compare the effect of Phyllantus versus placebo on profile of mood states (POMS) | 26 days
Compare the effect of Phyllantus versus placebo on cognitive performance tests | 26 days
  Using the CNS Vital Signs System
Compare the effect of Phyllantus versus placebo on sleep quality | 26 days
  Based on the number of hours slept

OTHER OUTCOMES:
Compare the effect of Phyllantus versus placebo on adverse events | 36 days
Compare the effect of Phyllantus versus placebo on a comprehensive metabolic panel (CMP) analysis | 26 days
Compare the effect of Phyllantus versus placebo on complete blood count | 26 days
Compare the effect of Phyllantus versus placebo on Urinalaysis | 26 days

CONTACTS AND LOCATIONS:
Overall Officials: Tengku Shahrir Tengku Adnan, Study Director — Biotropics Malaysia Berhad; Sanjay Udani, MD, Principal Investigator — Medicus Research, LLC
Locations (1):
- Medicus Research, LLC, Northridge, California, United States

IPD SHARING:
Plan to Share IPD: No